CLINICAL TRIAL: NCT07331818
Title: Luspatercept in Patients Affected With Rare Inherited Anemias
Acronym: LUSPARA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EuroBloodNet Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUSPARA - EuroBloodNet
Record Dates: First submitted 2025-12-05; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hereditary Red Blood Cell Disorder (Disorder)
MeSH Terms: interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LUSPATERCEPT (Experimental): All eligible subjects will receive a starting dose of luspatercept of 1 mg/kg on day
  1 of each 21 day cycle (every three weeks) In transfused patients, the first dose will be done at D8 from previous transfusion Responders at any dose will continue at the same dose until week 52 if they tolerate the drug (a follow up study will be envisaged)
  Interventions: Drug: Reblozyl

INTERVENTIONS:
Drug: Reblozyl — Reblozyl 25 mg powder for solution for injection / Reblozyl 75 mg powder for solution for injection

SUMMARY:
This is a prospective multicenter phase II basket trial evaluating Luspatercept in patients affected with rare inherited anemias

DETAILED DESCRIPTION:
This is a prospective multicenter phase II basket trial evaluating Luspatercept in patients affected with rare inherited anemias including : ✔ CSA group: constitutional non syndromic sideroblastic anemia () due to germline mutation including those with ALAS2, SLC25A38, SLC19A2, GLRX5, HSPA9. and other gene mutations ✔ CDA group: constitutional dyserythropïetic anemias ( (type I and II) ✔ NTD-DBA group: Diamond-Blackfan anemia (DBA) not requiring regular transfusion support (NTD-DBA) with or without continuous steroid therapy); (therapeutic independence or with continuous steroid therapy); 2 subgroups will be considered: RPS19 versus other genetic subgroups (RPL5, RPL11 and RPS26 mutations) ; to note these 4 genotypes account for the vast majority of patients

Patients will be recruited from centers of expertise within the European Union (France and Italy). In total, 45 patients are will be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Patient affected with a rare constitutional anemia including. :

   * constitutional non syndromic sideroblastic anemia (CSA) including those due to germline mutation in ALAS2, SLC25A38, SLC19A2, GLRX5, HSPA9 and also more rare cases with other mutations. . Patients without genetic diagnosis (currently up to 30% of CSa patients may be included after approval of PI and geneticists
   * constitutional dyserythropïetic anemias CDA (type I and II)
   * Diamond-Blackfan anemia not requiring regular transfusion support (NTD-DBA) (therapeutic independence or with continuous steroid therapy); 2 subgroups should be considered: RPS19 versus other genetic subgroups (mainly RPL5, RPL11 and RPS26 variants). Inclusions will be considered in order to have at least 3 patients in each subgroup before to expand inclusions
2. For diseases of the three subtypes (CSA, CDA, and DBA-NTD), diagnosis must be supported genetically by presence of ACMG class 4 or 5 variant(s).
3. Age ≥18 years at the first screening
4. For CSA and CDA, both Transfusion dependent (TD) patients and Non Transfusion dependent (TD) patients may be included:

   * TD patients: transfusion-dependency definition is: 6 to 20 units of packed red cells within previous 24 weeks with no transfusion-free period of > 56 days (except for DBA patients for whom transfusion dependency is a factor of exclusion)
   * NTD patients: patients must have significant anemia e.g. hemoglobin < 10.5 gr/dl (average of at least 2 Hb measurements separated by a minimum of 7 days during screening period) occasional transfusion aloowed if ≤ 5 red-cell units per 24 weeks and red blood cell transfusion free > 8 weeks before inclusion
5. Adequate renal function, defined by creatinine less than 1.5 times the upper limit of normal, creatinine clearance ≥ 30 mL/min (MDRD formula).
6. Adequate liver function, defined by transaminases and gamma-glutamyl transferase less than 1.5 times the upper limit of normal.
7. ECOG performance status 0-2 at the time of screening.
8. Be willing and able to give written informed consent and to comply to all study procedures for the duration of the study.
9. A FCBP (female of childbearing potential) for this study was defined as a sexually mature woman who: (1) had not undergone a hysterectomy or bilateral oophorectomy; or (2) had not been naturally postmenopausal (amenorrhea following cancer therapy did not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months). A FCBP participating in the study must:

   * Have had 2 negative pregnancy tests as verified by the investigator prior to starting the Investigational Product (IP) (unless the screening pregnancy test was done within 72 hours of Cycle 1 Day 1). She must have had agreed to ongoing a monthly pregnancy testing during the course of the study and after EOT
   * If sexually active, agreed to have used, and been able to comply with, highly effective contraception** without interruption, 5 weeks prior to starting IP, during treatment with IP (including dose interruptions), and for 12 weeks after discontinuation of IP. ** Highly effective contraception was defined in this protocol as the following (information also appeared in the ICF): Hormonal contraception (eg, birth control pills, injection, implant, transdermal patch, vaginal ring), intrauterine device, tubal ligation (tying your tubes), or a partner with a vasectomy
10. Male subjects must: Have agreed to use a condom, defined as a male latex condom or nonlatex condom NOT made out of natural (animal) membrane (eg, polyurethane), during sexual contact with a pregnant female or a FCBP while participating in the study, during dose interruptions, and for at least 12 weeks following IP discontinuation, even if he had undergone a successful vasectomy

Exclusion Criteria:

1. DBA patients with transfusion dependency or DBA patients with non RPS19, RPS26, RPL5 or RPL11 genotype or without gene identification
2. For patients with CSA and no established genetic diagnosis, acquired sideroblastic anemia and SF3B1 variant should be excluded with non RPS19, RPS26, RPL5 or RPL11 genotype or without gene identification
3. Severe infection or any other uncontrolled severe condition.
4. Uncontrolled hypertension
5. Significant cardiac disease - NYHA Class III or IV or having suffered a myocardial infarction in the last 6 months.
6. Use of investigational agents within 30 days or any anticancer therapy (including IMiD) within 2 weeks before the study entry. The patient must have recovered at least a grade 1 from all acute toxicity from any previous therapy.
7. Use of EPO within 4 weeks of study entry
8. Active cancer or cancer during the year prior to trial entry other than basal cell carcinoma, or carcinoma in situ of the cervix or breast.
9. Patient already enrolled in another therapeutic trial of an investigational drug.
10. Known HIV infection or active hepatitis B or C.
11. Women who are or could become pregnant or who are currently breastfeeding.
12. Any medical or psychiatric contraindication that would prevent the patient from understanding and signing the informed consent form.
13. Patient eligible at short or medium term for allogeneic stem cell transplantation.
14. Known allergies to luspatercept or any of its excipients.
15. No affiliation to a health insurance system
16. For men and women of reproductive potential: unwillingness to be abstinent or use double anticonception during the trial period.
17. Persons deprived of liberty by judicial or administrative decision
18. Persons subject to a legal protection measure (guardianship, curatorship, safeguard of justice)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluating Luspatercept in patients affected with rare inherited anemias - Transfusion dependent patients | Up to 52 weeks
  the proportion of patients who achieve an erythroid response, defined as a reduction in the transfusion burden of at least 33% from baseline (the 12-week period before the first dose of luspatercept) during 12 weeks plus a reduction of at least 2 red cell units over this 12-week interval.
Evaluating Luspatercept in patients affected with rare inherited anemias - Non Transfusion dependent patients | Up to 52 weeks
  the proportion of patients with a mean hemoglobin concentration increase of 1.0 g/dL or higher from baseline over a continuous 12-week interval in the absence of red blood cell transfusions

SECONDARY OUTCOMES:
Proportion of Transfusion dependent patients with a reduction in the transfusion burden (33 % / week 13 - 24) | UP to 52 weeks
  Proportion of patients with a reduction in the transfusion burden of at least 33% from baseline during weeks 13 through 24 plus a reduction of at least 2 red-cell units over this 12-week interval
Proportion of Transfusion dependent patients with a reduction in the transfusion burden (50% / week 13 - 24) | UP to 52 weeks
  Proportion of patients with a reduction in the transfusion burden of at least 50% from baseline during weeks 13 through 24 plus a reduction of at least 2 red-cell units over this 12-week interval
Proportion of Transfusion dependent patients with a reduction in the transfusion burden (33 % / week 37 - 48) | UP to 52 weeks
  Proportion of patients with a reduction in the transfusion burden of at least 33% from baseline during weeks 37 through 48 plus a reduction of at least 2 red-cell units over this 12-week interval,
Proportion of Transfusion dependent patients with a reduction in the transfusion burden (50 % / week 37 - 48) | UP to 52 weeks
  Proportion of patients with a reduction in the transfusion burden of at least 50% from baseline during weeks 37 through 48 plus a reduction of at least 2 red-cell units over this 12-week interval
mean change from baseline in the transfusion burden | UP to 52 weeks
  mean change from baseline in the transfusion burden during weeks 13 through 24 and during weeks 37 through 48.
Proportion of Non Transfusion dependent patients - hemoglobin concentration | UP to 52 weeks
  mean change from baseline in hemoglobin concentration over a continuous 12-week interval (weeks 13-24)
Proportion of Non Transfusion dependent patients - hemoglobin concentration increase | UP to 52 weeks
  Proportion of Non Transfusion dependent patients with a mean hemoglobin concentration increase of 1.5 g/dL or higher from baseline over a continuous 12-week interval (weeks 13-24 and weeks 37-48) in the absence of red blood cell transfusions
Proportion of Non Transfusion dependent patients - duration of mean hemoglobin concentration | UP to 52 weeks
  Proportion of Non Transfusion dependent patients - duration of mean hemoglobin concentration increase of 1.0 g/dL or higher from baseline"

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Leblanc, Phd, Principal Investigator — Assistance Publique Hôpitaux de Paris - Hôpital Robert-Debré
Locations (6):
- France (5):
  - GCS Groupement des Hôpitaux de l'Institut Catholique de Lille, Lille
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Assistance Publique Hôpitaux de Paris - Hôpital Saint-Louis, Paris
  - Assistance Publique Hôpitaux de Paris - Hôpital Necker, Paris
  - CHU Bordeaux-Hôpital Haut-Lévêque, Pessac
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No